CLINICAL TRIAL: NCT05147987
Title: Improving Lactation Success in Black Mothers of Critically Ill Infants in the NICU Using Discreet, Hands-free, Wearable Breast Pumps
Brief Title: Improving Lactation Success in Black Mothers of Critically Ill Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202102029
Record Dates: First submitted 2021-11-08; First posted 2021-12-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2024-11

CONDITIONS: Insufficient Lactation
MeSH Terms: conditions — Lactation Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Will be provided a discreet, hands-free, wearable breast pump with an associated App
  Interventions: Device: Hands free wearable breast pump
- Standard care group (No Intervention): Will be provided a standard mechanical breast pump with no associated App.

INTERVENTIONS:
Device: Hands free wearable breast pump — Use of a supplementary breast pump which can be discreetly worn and is hands free
  Arms: Intervention Group

SUMMARY:
Racial disparities result in Black infants in the neonatal intensive care unit (NICU) receiving less breast milk (BM) than White and Hispanic infants.1 BM improves infant health yet mothers of critically ill infants produce insufficient amounts to provide these benefits which is likely due to inadequate daily breast pumping frequency. Black mothers face unique challenges to frequent breast pumping including returning to work earlier, working in facilities with inadequate lactation support, and limited privacy for breast pumping at home. Therefore, the objective of this pilot study is to determine the feasibility and potential benefits of using a discreet, hands-free, wearable breast pump with an associated App that tracks pumping frequency and BM production to increase lactation success in Black mothers of infants admitted to the NICU. Specific aims include (1) evaluate the feasibility of a discreet, hands-free, wearable pump in Black mothers of critically ill infants to increase pumping frequency and BM production and (2) assess whether results indicate a signal of effectiveness supporting a subsequent adequately powered randomized clinical trial (RCT). Following delivery, 40 Black mothers of critically ill infants will be randomized to one of two groups. Group 1 will be provided a discreet, hands-free, wearable breast pump with an associated App and Group 2 will be provided a standard mechanical breast pump with no associated App. Results will be used to revise the intervention and study processes and to estimate outcome measurement variability and effect sizes needed for sample size calculations for an adequately powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* Mothers self-identified as Black
* > 18 years of age
* English speaking
* Stated intent to provide breast milk to her infant
* Rate their level of commitment to pumping breast milk for their infant for at least 3 weeks as 3 or greater or a 1-5 point Likert scale
* State they are available for an approximately 30 minute education session prior to hospital discharge
* Infant not expected to be stable enough to bottle/breastfeed for > 21 days
* Access to a mobile phone and able to download app.

Exclusion Criteria:

* Known illicit drug use
* Breast reduction or augmentation
* Positive HIV status
* Infant not expected to live > 7 days following delivery
* Has pacemaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants acceptance of the intervention | at 20-22 days
  Survey questions regarding the number of participant acceptance of intervention

SECONDARY OUTCOMES:
Expressed milk volume | up to 21 days
  Volume of expressed milk volume
Time to secretory activation | Up to 7 days
  Time from birth to expression of at least 20 mL of milk in 2 consecutive expressions
Expression frequency | up to 21 days
  How often mothers express daily
Lactation duration | up to 100 days
  how long mothers continue lactating
Infant consumption | up to 100 days
  percentage of feedings consisting of mother's milk consumed by infants

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parker, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No